CLINICAL TRIAL: NCT05119088
Title: Development of a Test Battery for Measurement of Knee Function in Patients With Patellar Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haraldsplass Deaconess Hospital (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Trine Hysing-Dahl, Principal Investigator, Haraldsplass Deaconess Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 185067
Record Dates: First submitted 2021-10-05; First posted 2021-11-12 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Patella; Joint Instability; Patellofemoral Joint Dislocation
MeSH Terms: conditions — Patella Fracture; Joint Instability; Patellar Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Return to Sport testbattery — At baseline, approximately 3 weeks before surgery and 6 months after surgery: patients conduct a testbattery consisting of 2 PROMs: the NPI-No and BPII2.0-No together with three physical tests: isokinetic strength tests, hop tests and Y-balance test. For the cross-cultural validation of NPI and BPII2.0 patients also conduct KOOS, IKDC 2000 and Tampa Scale.
  Other Names: Validation of Banff Patellofemoral Instability Instrument 2.0 - No; Validation of Norwich Instability Score - No

SUMMARY:
About six months after patella stabilizing surgery postoperative restrictions are commonly lifted and patients may consider whether a return to activity/sports is feasible. Currently, there are no evidence-based criteria to determine a patients readiness for sports and/or activity (RTS) following stabilizing surgery. The purpose of this project was therefore to investigate the feasibility of a test battery to evaluate knee function in postoperative follow-up evaluation - and in RTS decisions - for patients with patellar instability. Banff Patellofemoral Instability Instrument 2.0 and Norwich Patellar Instability Score is being translated and validatend in a Norwegian population. Furter is patients experience of living with patellar instability explored.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone surgical treatment for recurrent patellar dislocation in Helse Vest. The investigators will include patients with reconstruction of the medial patella femoral ligament, trochleaplasty, tibial tubercle osteotomy, Insall or concomitant procedures.

Exclusion Criteria:

* Unable to give written informed consent.
* Medial patellar dislocation.
* unable to understand written or spoken Norwegian.
* patients with other knee injuries.

Ages: 13 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Banff Patellofemoral Instability Instrument 2.0 change from pre- to postopertaive score | Baseline and 6 months after surgery.
  Self-administered, disease-specific quality of life score. It will be administered as a patient completed questionnaire.
Norwich patellar Instability score change from pre- to postopertaive score. | Baseline and 6 months after surgery.
  Patient-perceived symptoms of patellar instability during activity. It will be administered as a patient completed questionnaire.

SECONDARY OUTCOMES:
Y-balance test | Baseline and 6 months after surgery.
  Evaluates knee stability and asymmetrical balance in three directions (anterior, posteromedial and posterolateral).
Single legged hop tests | Baseline and 6 months after surgery.
  Comprises four tasks: single-leg hop for distance, triple hop for distance, triple cross-over hop for distance and six-meter timed hop.
Isokinetic strength test | Baseline and 6 months after surgery.
  Strength testing of knee extension / flexion (Biodex system 4 dynamometer, Biodex Medical Systems Inc., Shirley, New York). With a standardized protocol of five repetitions at 60 o/sec and 30 repetitions at 240 o/sec.
IKDC-2000 | Baseline and 6 months after surgery.
  Is a knee-specific, patient reported tool, including 18 questions across three domains: symptoms, physical activity and function. It will be administered as a patient completed questionnaire.
KOOS | Baseline and 6 months after surgery.
  Is an instrument to assess the patient's opinion about their knee and associated problems. It comprises five domains: pain, other symptoms, function in daily living, function in sports and recreational activities and knee-related QOL. It will be administered as a patient completed questionnaire.
Tampa scale of kinesiophobia | Baseline and 6 months after surgery.
  TSK is a 17-item patient-reported questionnaire aimed at quantifying the fear of re-injuries due to movement and physical activity. It will be administered as a patient completed questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Haraldsplass Deaconess Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hysing-Dahl T, Magnussen LH, Faleide AGH, Inderhaug E. Feasibility of return to sports assessment 6 months after patellar instability surgery. BMC Musculoskelet Disord. 2023 Aug 18;24(1):662. doi: 10.1186/s12891-023-06767-2. PMID 37596551
- [Derived] Hysing-Dahl T, Inderhaug E, Faleide AGH, Magnussen LH. Patients' experiences of living with patellar instability before and after surgery: a qualitative interview study. BMJ Open. 2023 Jun 9;13(6):e072141. doi: 10.1136/bmjopen-2023-072141. PMID 37295823